CLINICAL TRIAL: NCT02039401
Title: A Phase I/II, Open Label Study to Assess the Safety and Tolerability of VM202 in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Safety Study of VM202 to Treat Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMALS-001 / B
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's disease; neurodegenerative disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VM202 (Experimental): Total dose of 64 mg of VM202 It will be administered over the course of four visits: Day 0, Day 7, Day 14, and Day 21. As in all previous VM202 studies, final dose of VM202 for each target muscle group is divided and administered 2 weeks apart.
  Interventions: Biological: VM202

INTERVENTIONS:
Biological: VM202

SUMMARY:
The purpose of this study is to determine the safety and tolerability of intramuscular injections of VM202 at different injection sites in people with amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
A phase I/II, open label, single center study designed to assess the safety and tolerability of intramuscular injections of VM202 inpatients with Amyotrophic Lateral Sclerosis. Study enrollment will be staged. Enrollment will be halted after the sixth subject qualifies for treatment. A Data Safety Monitoring Board will conduct a safety evaluation after the first patient treated completes the Day 60 follow-up evaluation and the five other sequentially enrolled subjects complete at least the Day 30 follow-up. Enrollment will be suspended until a formal recommendation to proceed (or not proceed) is made by the Data Safety Monitoring Board.

Patients aged ≥ 21 years, but ≤ 75 years diagnosed with clinically definite, clinically probable, or clinically probable-laboratory supported Amyotrophic Lateral Sclerosis.

This study is not powered to detect differences in efficacy measures. However, descriptive statistics (N, mean, median, standard deviation, minimum and maximum values, where applicable) of clinically meaningful endpoints will be tabulated

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years, but < or = 75 years
* Subjects diagnosed with:

  * clinically definite Amyotrophic Lateral Sclerosis,
  * clinically probable Amyotrophic Lateral Sclerosis, or
  * clinically probable-laboratory supported Amyotrophic Lateral Sclerosis as specified in the revised El Escorial / Airlie House diagnostic criteria
* Onset of ALS < 2 years at Screening
* Forced Vital Capacity ≥ 60% of predicted
* Revised Amyotrophic Lateral Sclerosis Functional Rating Scale ≥ 30
* Not taking riluzole, or on a stable dose for at least thirty days prior to Screening (defined as no noted toxicities)
* Able and willing to give informed consent
* If female of childbearing potential, negative urine pregnancy test at Screening and using acceptable method of birth control during the study.

Exclusion Criteria:

* Neurological symptom(s) due to vitamin B12 deficiency
* Requires tracheotomy ventilation or noninvasive ventilation > 16 hours / day
* Comorbidities such as Parkinson's disease, schizophrenia, renal failure, or any other severe complication that, in the Investigator's opinion, will compromise the safety of the patient or confound interpretation of the data collected in this study
* Other neuromuscular disease
* Inflammatory disorder of the blood vessels (inflammatory angiopathy, such as Buerger's disease)
* Active infection
* Chronic inflammatory disease (e.g., Crohn's disease, rheumatoid arthritis)
* Positive HIV or HTLV at Screening
* Active Hepatitis B or C as determined by Hepatitis B core antibody, antibody to Hepatitis B surface antigen (IgG and IgM), Hepatitis B surface antigen and Hepatitis C antibodies at Screening
* Subjects with known immunosuppression or currently receiving immunosuppressive drugs, chemotherapy or radiation therapy
* Stroke or myocardial infarction within last 3 months
* Patients with a recent history (< 5 years) of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence);
* Subjects requiring > 81 mg daily of acetylsalicylic acid; subjects may be enrolled if willing/able to switch to ≤ 81 mg daily of acetylsalicylic acid or to another medication
* Subjects requiring regular COX-2 inhibitor drug(s) or non-specific COX-1/COX-2 inhibiting drugs, or high dose steroids (excepting inhaled steroids); subjects may be enrolled if willing/able to undergo medication wash-out prior to the first dosing and to refrain from taking these drugs for the duration of the study
* Have used an investigational drug within 30 days of Screening
* Pregnant or currently lactating
* Major psychiatric disorder in past 6 months
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the Investigator are not suitable to participate.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2015-08-03 (Actual); Study Completion 2024-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Kessler, MD, Principal Investigator — Northwestern University Stem Cell Institute
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sufit RL, Ajroud-Driss S, Casey P, Kessler JA. Open label study to assess the safety of VM202 in subjects with amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017 May;18(3-4):269-278. doi: 10.1080/21678421.2016.1259334. Epub 2017 Feb 6. PMID 28166654

RESULTS

PARTICIPANT FLOW:
Groups:
- Engensis (VM202) Group 1: Total dose of 64 mg of VM202, administered over the course of four visits: Day 0, Day 7, Day 14, and Day 21. As in all previous VM202 studies, final dose of VM202 for each target muscle group is divided and administered 2 weeks apart. Group 1 received Engensis IM injections beginning with the lower limbs, with injection location (lower vs upper limbs) alternating weekly
  VM202
- Engensis (VM202) Group 2: Total dose of 64 mg of VM202, administered over the course of four visits: Day 0, Day 7, Day 14, and Day 21. As in all previous VM202 studies, final dose of VM202 for each target muscle group is divided and administered 2 weeks apart. Group 2 received Engensis IM injections beginning with the upper limbs, with injection location (lower vs upper limbs) alternating weekly
  VM202
Period: Overall Study
Arm/Group | Engensis (VM202) Group 1 | Engensis (VM202) Group 2
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Engensis (VM202) Group 1 | Engensis (VM202) Group 2 | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.9) | 55.8 (3.0) | 52.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious and Non Serious Adverse Events
Description: Adverse events (including serious adverse events, and adverse events leading to treatment discontinuation) throughout the 9 months follow-up. Descriptive statistics will be used to characterize safety parameters.
Time Frame: Throughout the nine month follow up
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Total: All subjects in Groups 1 and 2
Arm/Group | Total
Number analyzed (Participants) | 18
Participants
  Diarrhoea | 1
  Gastroesophargeal reflux disease | 1
  Small intestinal obstruction | 1
  Asthenia | 1
  Fatigue | 1
  Pyrexia | 1
  Bronchitis | 1
  Eye infection | 1
  Lyme disease | 1
  Nasopharyngitis | 4
  Tooth abscess | 1
  Urinary tract infection | 1
  Fall | 11
  Muscle strain | 1
  Skin abrasion | 1
  Skin laceration | 2
  Blood pressure increased | 1
  Weight decreased | 1
  Arthralgia | 1
  Myalgia | 1
  Headache | 3
  Depression | 2
  Haematuria | 1
  Aspiration | 1
  Cough | 1
  Dyspnoea | 1
  Pneumonia aspiration | 1
  Respiratory failure | 1
  Respiratory tract congestion | 1
  Rash | 1

2. Secondary Outcome: The Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R)
Description: The Amyotrophic Lateral Sclerosis Function Rating Scale includes twelve questions that ask the physician to rate his/her impression of the patient's level of functional impairment in performing one of twelve common tasks (e.g., climbing stairs). Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0 = worst and 48 = best.
Time Frame: Screening, on Day 0 before the treatment (injection), on Day 30, Day 60, Day 90, at 6 months and 9 months
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Overall: Total subjects from Groups 1 and 2
Arm/Group | Engensis (VM202) Group 1 | Engensis (VM202) Group 2 | Overall
Number analyzed (Participants) | 9 | 9 | 18
units on a scale
  Screening | 39.89 (3.26) | 38.11 (4.62) | 39 (3.99)
  Day 0 | 40.22 (2.99) | 37.11 (5.25) | 38.67 (4.45)
  Day 30 | 40 (3.94) | 35 (6.44) | 37.5 (5.78)
  Day 60 | 39.25 (3.65) | 33.44 (6.46) | 36.18 (5.97)
  Day 90 | 38.22 (3.11) | 33.89 (6.05) | 36.06 (5.17)
  Month 6 | 35.5 (4.5) | 29.25 (8.5) | 32.38 (7.32)
  Month 9 | 31.22 (4.97) | 25.88 (8.51) | 28.71 (7.18)

3. Secondary Outcome: Change in Mean Muscle Strength Medical Research Council (MRC) Scores
Description: The Medical Research Council (MRC) Scale is a validated instrument used in assessing muscle strength. It uses the numeral grades 0-5 to characterize muscle strength as follows: 0 - No contraction;1 - Flicker or trace contraction; 2 - Active movement, with gravity eliminated; 3 - Active movement against gravity; 4 - Active movement against gravity and resistance; 5 - Normal power The MRC scale was used to assess muscle strength in the muscle groups injected with Engensis.
Time Frame: Day 0, Day 30, Day 60, Day 90, at 6 months and 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis (VM202) Group 1 | Engensis (VM202) Group 2 | Overall
Number analyzed (Participants) | 9 | 9 | 18
score on a scale
  Day 30 | -0.67 (3.54) | -3.78 (5.78) | -2.22 (4.92)
  Day 60 | -0.63 (3.81) | -2.89 (3.59) | -1.82 (3.76)
  Day 90 | -5.11 (4.7) | -4.56 (7.97) | -4.83 (6.35)
  Month 6 | -8.25 (5.2) | -13.63 (7.25) | -10.94 (6.7)
  Month 9 | -17.38 (11.39) | -18.63 (10.03) | -18.0 (10.39)

4. Secondary Outcome: Change From Baseline (Day 0) in Forced Vital Capacity (%)
Description: pulmonary function test that quantifies the volume of air that can forcibly be blown out after full inspiration. It correlates with survival in ALS
Time Frame: Day 30, Day 60, Day 90, at 6 months and 9 months
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Engensis (VM202) Group 1 | Engensis (VM202) Group 2 | Overall
Number analyzed (Participants) | 9 | 9 | 18
percentage
  Day 30 | -1.67 (5.12) | -4.11 (6.15) | -2.89 (5.63)
  Day 60 | -5 (7.03) | -8.33 (10.3) | -6.76 (8.81)
  Day 90 | -8 (7.5) | -13.44 (12.45) | -10.72 (10.36)
  Month 6 | -11.13 (9.76) | -24 (22.17) | -17.56 (17.84)
  Month 9 | -16.63 (11.83) | -29.88 (18.78) | -23.25 (16.64)

ADVERSE EVENTS:
Time Frame: Day 0 through the Month 9 visit
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=18)
small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=18)
diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4)
Tooth abscess (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 11 (21)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Skin abraision (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Blood pressure increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT02039401/Prot_SAP_000.pdf